CLINICAL TRIAL: NCT04404907
Title: Analysis of Tanning Attitudes and Behaviors by Young Adult Sexual Minority Males in the Greater Chicago Area
Brief Title: Deliberate Ultraviolet Light Exposure to Get a Tan by Young Adult Sexual Minority Males
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Research Professor of Dermatology, Northwestern University
Other Study IDs: STU00206314
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Sun Sensitivity
MeSH Terms: conditions — Photosensitivity Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males who never deliberately tan: Males responded to an anonymous online survey that they never deliberately tan
  Interventions: Other: no intervention
- Males who ever deliberately tan: Males responded to an anonymous online survey that they had ever deliberately tan
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is a secondary analysis of registry data.

SUMMARY:
The purpose of this study is to: a) identify enablers and barriers to deliberate ultraviolet light exposure by young sexual minority men (SMM), and b) quantify the extent of their deliberate ultraviolet light exposure.

DETAILED DESCRIPTION:
Aim 1: To develop survey items to assess tanning attitudes and behaviors Nine survey items used by the PI in previous deliberate tanning research were adapted with the expert consensus of members of Northwestern's Institute for Sexual and Gender Minority Health and Wellbeing. Discussions with the PI, research personnel and members of the institute developed the hypothesis that in addition to the previously reported appearance motivations young SMM may be engaging in tanning (indoors or outdoors) as a social activity. A tenth survey item was developed to assess deliberate tanning as a social activity.

Aim 2: Analyze the tanning attitudes and behavior data acquired in an online survey of young adult sexual minority males, who regularly participate in the RADAR study.

RADAR is a longitudinal study with cohorts from the greater Chicago region recruited between 2008 and 2015. The 10 survey items about tanning attitudes and behaviors were added to the online survey that examines SMMs' behavior in the prior 6 months. This is a secondary analysis of registry data acquired by the RADAR study.

ELIGIBILITY:
Inclusion Criteria:

* Young adult SMM (age 18-39)
* Able to read English
* Have internet access
* Willing to complete the online survey

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes — Participants self-identify as sexual minority males
Study Population: RADAR is a longitudinal study with cohorts from the greater Chicago region recruited between 2008 and 2015. Participants respond to online surveys every 6 months.
Sampling Method: Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Since all data is deidentified, the results cannot be shared individually; however, the results may be provided to the entire cohort in a newsletter.

REFERENCES:
- [Result] Robinson JK, Wahood S, Stapleton JL. Motives for intentional sunlight exposure among young adult sexual minority men: appearance, relaxation and socialization in a cohort study. Br J Dermatol. 2021 Mar;184(3):563-564. doi: 10.1111/bjd.19609. Epub 2020 Nov 18. No abstract available. PMID 33067803
- Available data/document: Clinical Study Report — http://doi.org/10.3886/ICPSR37603.v1 — Mustanski, Brian. Multilevel Influences on HIV and Substance Use in a YMSM Cohort (RADAR) - Visit #1, Chicago Metropolitan Area, 2015-2018. Inter-university Consortium for Political and Social Research [distributor], 2020-03-19.

RESULTS

PARTICIPANT FLOW:
Groups:
- Males Who Never Deliberately Tan: Registry survey of males responded with a history of never deliberately (intentionallly) tanned
- Males Who Ever Deliberately Tanned: Registry survey of males responded with a history of ever deliberately (intentionallly) tanned to make their skin appear darker
Period: Overall Study
Arm/Group | Males Who Never Deliberately Tan | Males Who Ever Deliberately Tanned
Started | 442 | 95
Occasional Tan (2-10 times in 3 months) | 0 | 88
Frequent Tan (>10 times in 3 months) | 0 | 7
Completed | 442 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Males Who Never Deliberately Tan | Males Who Ever Deliberately Tanned | Total
Number analyzed (Participants) | 442 | 95 | 537
Age, Continuous [Mean (Standard Deviation); unit: years] — REDCap survey online
  years | 24.71 (3.2) | 24.14 (2.8) | 24.42 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 442 | 95 | 537
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 136 | 41 | 177
  Not Hispanic or Latino | 306 | 54 | 360
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 15 | 2 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 171 | 9 | 180
  White | 221 | 75 | 296
  More than one race | 31 | 9 | 40
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 442 | 95 | 537
Highest level of education [Count of Participants; unit: Participants]
  high school or less | 108 | 14 | 122
  trade school | 12 | 4 | 16
  some college | 189 | 32 | 221
  college graduate | 94 | 38 | 132
  some graduate school | 19 | 6 | 25
  graduate degree | 20 | 1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Outdoor Tanning Motives
Description: The 95 participants who self-reported deliberate tanning responded to 7 online survey items reported in the analysis population description.
Time Frame: 14 days
Population: Responses to 7 survey items using Likert scale [1= strongly disagree (not at all concerned), 3= neither agree nor disagree, 5= strongly agree (extremely concerned)] were entered online
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Occasional Tanning: Males who deliberately (intentionally tanned) 2-10 times in 3 months
- Frequent Tanning: Males who intentionally tanned 10 or more times in 3 months
Arm/Group | Occasional Tanning | Frequent Tanning
Number analyzed (Participants) | 88 | 7
score on a scale
  Most other gay and bisexual guys like me feel more attractive with a tan | 3.64 (1.01) | 3.81 (1.05)
  Tanning helps me relax | 4.10 (0.78) | 4.29 (0.70)
  Feel more confident with a tan | 3.09 (0.80) | 3.03 (1.13)
  Go tanning with others as a social activity | 4.09 (0.80) | 4.55 (0.31)
  Important to protect skin from the sun | 3.07 (0.73) | 3.00 (1.10)
  Concern about skin cancer | 2.86 (0.86) | 3.00 (1.41)
  Chance of getting skin cancer is high | 3.01 (0.88) | 3.07 (1.50)
Statistical Analysis 1: Comparison: Occasional Tanning vs Frequent Tanning; feel more attractive; Test type: Other — ANOVA; p = 0.02, ANOVA
Statistical Analysis 2: Comparison: Occasional Tanning vs Frequent Tanning; tanning helps relax; Test type: Other — ANOVA; p = 0.001, ANOVA
Statistical Analysis 3: Comparison: Occasional Tanning vs Frequent Tanning; confident with a tan; Test type: Other; p = 0.34, ANOVA
Statistical Analysis 4: Comparison: Occasional Tanning vs Frequent Tanning; Social activity; Test type: Other; p = 0.0004, ANOVA
Statistical Analysis 5: Comparison: Occasional Tanning vs Frequent Tanning; Important to protect skin from the sun; Test type: Other; p = 0.66, ANOVA
Statistical Analysis 6: Comparison: Occasional Tanning vs Frequent Tanning; Concern about develop skin cancer; Test type: Other; p = 0.16, ANOVA
Statistical Analysis 7: Comparison: Occasional Tanning vs Frequent Tanning; Chances of getting skin cancer are high; Test type: Other; p = 0.29, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Males Who Never Deliberately Tan; Males Who Ever Deliberately Tanned: No adverse events reported in the online survey of this group
Arm/Group | Males Who Never Deliberately Tan | Males Who Ever Deliberately Tanned
All-Cause Mortality (participants affected / at risk) | 0/442 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/442 | 0/95
Other Adverse Events (participants affected / at risk) | 0/442 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04404907/Prot_SAP_000.pdf